CLINICAL TRIAL: NCT04543968
Title: Open Label Pilot Study Using Hydroxytyrosol (HT) as a Dietary Supplement in Patients With Mitochondrial Diseases (MDs)
Brief Title: Clinical Study of Hydroxytyrosol (HT) in Mitochondrial Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Children's Hospital (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fung Cheuk Wing, Consultant, Hong Kong Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Clinical study of HT in MDs
Record Dates: First submitted 2020-07-31; First posted 2020-09-10 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Mitochondrial Diseases
Keywords: mitochondria; mitochondrial diseases; MD; mitochondrial dysfunction; mitochondrial respiratory chain; MRC; oxidative phosphorylation; OXPHOS; mitochondrial
MeSH Terms: conditions — Mitochondrial Diseases | interventions — 3,4-dihydroxyphenylethanol

STUDY DESIGN:
Intervention Model Description: Twelve subjects will be recruited, including MD patients with confirmed MD-associated nuclear DNA or mtDNA mutations. Subjects will receive hydroxytyrosol (HT) daily as dietary supplements for 12 months. After that, patients will be randomly assigned in 1:1 ratio to either continue on or withdraw from receiving hydroxytyrosol (HT) as their dietary supplements for another 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydroxytyrosol (HT) intake (Experimental): MD patients will receive hydroxytyrosol (HT) daily as dietary supplements for 12 months. After that, patients will be randomly assigned in 1:1 ratio to continue on receiving hydroxytyrosol (HT) as their dietary supplements for another 6 months.
  Doses of hydroxytyrosol (HT) intake: (1) 3-10 years old, 10 mg/day; (2) 11-18 years old 30mg/day
  Interventions: Dietary Supplement: hydroxytyrosol (HT) intake
- hydroxytyrosol (HT) intake and withdraw (Experimental): MD patients will receive hydroxytyrosol (HT) daily as dietary supplements for 12 months. After that, patients will be randomly assigned in 1:1 ratio to withdraw from receiving hydroxytyrosol (HT) as their dietary supplements for another 6 months.
  Doses of hydroxytyrosol (HT) intake: (1) 3-10 years old, 10 mg/day; (2) 11-18 years old 30mg/day
  Interventions: Dietary Supplement: hydroxytyrosol (HT) intake and withdraw

INTERVENTIONS:
Dietary Supplement: hydroxytyrosol (HT) intake — MD patients will receive hydroxytyrosol (HT) daily as dietary supplements for 12 months. After that, patients will be randomly assigned in 1:1 ratio to continue on receiving hydroxytyrosol (HT) as their dietary supplements for another 6 months.
  Arms: hydroxytyrosol (HT) intake
Dietary Supplement: hydroxytyrosol (HT) intake and withdraw — MD patients will receive hydroxytyrosol (HT) daily as dietary supplements for 12 months. After that, patients will be randomly assigned in 1:1 ratio to withdraw from receiving hydroxytyrosol (HT) as their dietary supplements for another 6 months.
  Arms: hydroxytyrosol (HT) intake and withdraw

SUMMARY:
Mitochondrial diseases (MDs) are the commonest group of inborn errors resulting from primary dysfunction of mitochondrial respiratory chain (MRC). High phenolics-containing extra-virgin olive oil (EVOO) can be one of the potential dietary supplements for the treatment of MD. Previous reports demonstrated that phenolics including oleuropein, oleocanthal, hydroxytyrosol and tyrosol found in EVOO have strong antioxidant properties against the oxidative stress in brain tissue and showed a protective effect on mitochondria by restoring mitochondrial enzymatic activities.

This proposed study is an open-label pilot/ feasibility clinical trial using hydroxytyrosol (HT) as dietary supplements in a cohort of 12 MD patients recruited from the Hong Kong Children's Hospital (HKCH).

The objective is to explore the longitudinal effect of receiving hydroxytyrosol (HT) as dietary supplements over a 12-month period and the change on a 6-month period after withdrawal. The applicability of the outcome measures will be evaluated in the current trial for future clinical studies and obtain relevant data for the next phase of the clinical trial on hydroxytyrosol (HT) efficacy. Besides, the tolerability of hydroxytyrosol (HT) in MD patients will be evaluated.

The primary outcome measure is the functional assessment of the patient's clinical outcomes by International Paediatric Mitochondrial Disease Score (IPMDS). Secondary outcome measures included the measurement of biochemical and radiological parameters. Besides, tolerability and quality of life of the subjects will be determined.

Relevant data including the feasibility of subject recruitment, withdrawal rate, feasibility of data collection of outcome measures, longitudinal effect of hydroxytyrosol (HT) on the outcome measures in the trial can be collected and analysed in this pilot study providing important information for the future clinical trials. The ultimate goal is to develop effective therapies to lower mortality, improve the clinical outcomes and quality of life in MD patients.

DETAILED DESCRIPTION:
High phenolics-containing extra-virgin olive oil (EVOO) can be one of the potential dietary supplements for the treatment of MD. There is growing evidence to suggest that daily consumption of EVOO in Mediterranean diets have beneficial effects on preventing neurodegeneration. Previous reports demonstrated that phenolics including oleuropein, oleocanthal, hydroxytyrosol and tyrosol found in EVOO have strong antioxidant properties against the oxidative stress in brain tissue and protective effect on both acute and chronic neurodegenerative diseases by in vitro study and animal models. In addition to improvement of arsenic-induced oxidative stress by oleuropein or hydroxytyrosol treatment, hydroxytyrosol also showed a protective effect on mitochondria by restoring mitochondrial enzymatic activities in rat brain. In vitro study also demonstrated the stimulatory effect of hydroxytyrosol on mitochondrial function including in mouse 3T3-L1 adipocytes and human endothelial cells. A recent reported clinical study showed that consumption of olive oil could increase mitochondrial membrane fluidity and ATPase activity in patients with relapsing-remitting multiple sclerosis, a neurodegenerative disease associated with mitochondrial dysfunction.

Mitochondrial diseases (MDs) are the commonest group of inborn errors with a minimal prevalence of 12.5 per 100,000 and 4.7 per 100,000 adults and children respectively. These diseases are resulted from primary dysfunction of mitochondrial respiratory chain (MRC) which is mostly caused by both nuclear and mitochondrial DNA defects. They are progressive, multisystem disorders that can affect many parts of the body including brain, nerve, muscle, kidney, heart, liver, eyes, ears or pancreas and some are devastating or even life threatening. Development of effective treatments for the patients is an unmet need until now. Effective treatment strategies and clinical trials are limited, and therapies are mostly palliative. Drug developments and clinical trials for these diseases are scarce in Hong Kong when compared with other countries.

MDs are extremely heterogeneous phenotypically and genetically with the biochemical dysfunction and pathogenic mechanisms being unique in each individual molecular defect. With the advance in next generation sequencing, over 300 mitochondrial genes are implicated to cause human diseases. This wide heterogeneity has been hindering the development of new therapeutic strategies such as gene therapy which requires long term evaluation and substantial manipulation to improve efficacy and reduce toxicity risk. It is therefore not efficient nor realistic to develop unique therapy targeting at a specific molecular defect.

The future pharmaceutical development for treating mitochondrial dysfunctions will focus on boosting the residual mitochondrial function by non-specific bypassing the defective components of MRC or improving the aberrant cellular consequences. Dietary supplements were demonstrated to treat MD owing to their roles as metabolic cofactors to ameliorate mitochondrial ATP production, bypass mitochondrial complex defects and remove toxic metabolites. However, there are few randomized controlled trials to assess the cause-effect relationship of these dietary supplements.

The present study is a feasibility clinical trial to explore the longitudinal effect of receiving hydroxytyrosol (HT) as dietary supplements on primary and secondary outcomes (clinical, biochemical and radiological parameters and quality of life) and tolerability in MD patients in Hong Kong. The investigators aim to obtain relevant data to determine the sample size and treatment duration for the next phase of the clinical trial on hydroxytyrosol (HT) efficacy. Another aim of this study is to evaluate the applicability of the outcome measures in the current study for future clinical trials on different treatment strategies.

This pilot study will be a longitudinal, open label study. Twelve subjects will be recruited, including MD patients with confirmed MD-associated nuclear DNA or mtDNA mutations, from the Hong Kong Children's Hospital (HKCH). Subjects will receive hydroxytyrosol (HT) daily as dietary supplements for 12 months. After that, patients will be randomly assigned in 1:1 ratio to either continue on or withdraw from receiving hydroxytyrosol (HT) as their dietary supplements for another 6 months.

Hydroxytyrosol (HT) dosage are based on the past clinical trials in humans and the NOAEL. The willingness of the participants to stay in the trial in terms of the percentage of participants completing the whole trial on hydroxytyrosol (HT) dietary supplement will be assessed. The withdrawal rate in different study periods and the reasons of withdrawal will be further studied.

Subjects will visit the trial site at different time points after the start of dietary supplements for clinical follow up, functional assessment including questionnaire, blood and urine sampling and neuroimaging as primary and secondary outcome measures. There will be more frequent follow-up and monitoring after initiation and withdrawal of supplements. Data of primary and secondary outcome measures (except radiological evaluation) will be collected before the trial as baseline, 2 weeks, 6 weeks, 3, 6, 9, 12 months after the commencement of the trial and 2 weeks, 6 weeks, 3 and 6 months after randomization. The investigators will examine the feasibility of collecting data on the primary and secondary outcome measures in a clinical trial condition. The amount of missing data, the reason for the missing and difficulties on those data collection will be evaluated.

An open label trial is used for this proposed study because a matching placebo with the same properties, such as taste, smell, colour, etc, as hydroxytyrosol (HT) to keep blindness is not yet developed at this moment. Therefore, a withdrawal design will be used even though this can be a limitation of this study because of the easy accessibility of hydroxytyrosol (HT) by the patients who can continue to use EVOO on their own after being assigned for withdrawal, which may potentially affect the outcome. Information on any deviation from the study protocol on this issue can be collected from the patients by questionnaires at the end of the study to guide the data analysis and interpretation.

ELIGIBILITY:
Inclusion criteria

1. Subject (aged 3-18 years) is confirmed to have pathogenic MD-associated nuclear DNA or mtDNA mutations.
2. Subject is willing and able to comply with all requirements of the clinical trial.
3. Subject is given enough time and opportunity to consider his/her participation and has signed his/her written consent.

Exclusion criteria

1. Subject is participating or has participated within the last 2 months in any clinical trial involving hydroxytyrosol (HT) or hydroxytyrosol (HT) -associated phenols as dietary supplements.
2. Subject has a medical condition which can be exacerbated by hydroxytyrosol (HT) or hydroxytyrosol (HT) -associated phenols.
3. Subject has allergy to olive oil.
4. Subject is pregnant.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in International Paediatric Mitochondrial Disease Score | baseline, 2 weeks, 6 weeks, 3, 6, 9, 12 months after the commencement of the trial and 2 weeks, 6 weeks, 3 and 6 months after randomization
  International Paediatric Mitochondrial Disease Score was previously established by Radboud Centre for Mitochondrial Medicine to monitor symptoms and signs of disease progression in MD patients aged from 1-18 years old. This scale was suggested to be a robust tool for the follow-up of children with MD and aimed for the purpose in clinical trials. International Paediatric Mitochondrial Disease Score consists of 61 items in 3 domains (Domain 1, 2 and 3). Domain 1 has 23 items providing the detailed insights into subjective complaints and symptoms which should be assessed by interviewing parents or caregivers. Domain 2 consists of 25 items assessed by physical examination. Domain 3 has 13 items of functional assessment obtained by physical/motor function evaluation. Minimum value of raw score is 0 and maximum value is 243. Lower score means better clinical status.

SECONDARY OUTCOMES:
Change in blood gas parameter | Baseline, 2 weeks, 6 weeks, 3, 6, 9, 12 months after the commencement of the trial and 2 weeks, 6 weeks, 3 and 6 months after randomization
  Blood gases will be measured by electrochemical analysis which can reveal metabolic acidosis acting as one of the indicators for MD.
Change in plasma lactate/pyruvate ratio | Baseline, 2 weeks, 6 weeks, 3, 6, 9, 12 months after the commencement of the trial and 2 weeks, 6 weeks, 3 and 6 months after randomization
  Plasma lactate/ pyruvate will be measured by automated enzymatic method and marked elevation of plasma lactate/ pyruvate ratio suggests the presence of mitochondrial dysfunction because of a shift in mitochondrial redox state.
Change in plasma amino acid level | Baseline, 2 weeks, 6 weeks, 3, 6, 9, 12 months after the commencement of the trial and 2 weeks, 6 weeks, 3 and 6 months after randomization
  Plasma amino acids will be measured by liquid chromatography tandem mass spectrometry (LC-MS/MS). Increase in plasma amino acid level including alanine, glycine, proline and threonine will indicate an alteration of redox state caused by respiratory chain dysfunction.
Change in urine organic acid level | Baseline, 2 weeks, 6 weeks, 3, 6, 9, 12 months after the commencement of the trial and 2 weeks, 6 weeks, 3 and 6 months after randomization
  Urine organic acid will be measured by liquid chromatography tandem mass spectrometry (LC-MS/MS). Urine organic acid analysis can showed elevation of malate, fumarate, 3-methylglutaconic acid etc, in MD patients.
Change in Paediatric Quality Of Life assessment: Paediatric Quality of Life Inventory version 4.0 generic core scale | Baseline, 2 weeks, 6 weeks, 3, 6, 9, 12 months after the commencement of the trial and 2 weeks, 6 weeks, 3 and 6 months after randomization
  The measurement model the investigators will use will be the Paediatric Quality of Life Inventory version 4.0 generic core scale for the measurement of health-related quality of life in children and adolescents who are healthy or with acute and chronic health condition. Paediatric Quality Of Life assessment consists of 5 versions of the same questionnaire for various age ranges: a) toddler version for 2-4 year old; b) young child version for 5-7 years old; c) child version for 8-12 years old; d) adolescent version for 13-18 years old; e) young adult version for 18-23 years old. Each of the versions has a parent version for proxy report and child version for self-report (except for the toddler version). Each version is composed of 23 items with 4 scales (physical, emotional, social and school functioning) and 3 summary scores (total, physical health summary, psychosocial health summary score). The scale scores ranged from 0-100 and higher score indicates better quality of life.
Study of tolerability of hydroxytyrosol (HT): number of intervention-related adverse events | Baseline, 2 weeks, 6 weeks, 3, 6, 9, 12 months after the commencement of the trial and 2 weeks, 6 weeks, 3 and 6 months after randomization
  The MD patients will be followed up by a clinician during the time of functional assessment. The tolerability will be assessed by evaluating the number of intervention-related adverse events in patients taking hydroxytyrosol (HT) as dietary supplements. Adverse events were not reported in the literature but may potentially include gastrointestinal upset, vomiting, nausea, and diarrhea with subsequent weight loss.
Change in radiological evaluation | Baseline, 12 months after receiving hydroxytyrosol (HT) and 6 months after withdrawal or being maintained on hydroxytyrosol (HT) after randomization.
  Magnetic resonance imaging of the brain with spectroscopy will be used to evaluate patients' responses before the trial as baseline, 12 months after receiving EVOO and 6 months after withdrawal or being maintained on EVOO after randomization. Radboud Centre for Mitochondrial Medicine Pediatric MRI score (RCMM-PMRIS), will be used for the outcome measure. RCMM-PMRIS focuses on 6 most commonly described abnormalities in neuroimaging and define the extent of brain involvement. This can help to evaluate MD severity, disease progression and effect of treatment radiologically.

CONTACTS AND LOCATIONS:
Overall Officials: Cheuk Wing Fung, Principal Investigator — Hong Kong Children's Hospital
Locations (1):
- Hong Kong Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koene S, Hendriks JCM, Dirks I, de Boer L, de Vries MC, Janssen MCH, Smuts I, Fung CW, Wong VCN, de Coo IRFM, Vill K, Stendel C, Klopstock T, Falk MJ, McCormick EM, McFarland R, de Groot IJM, Smeitink JAM. International Paediatric Mitochondrial Disease Scale. J Inherit Metab Dis. 2016 Sep;39(5):705-712. doi: 10.1007/s10545-016-9948-7. Epub 2016 Jun 9. PMID 27277220
- [Background] Mancuso M, McFarland R, Klopstock T, Hirano M; consortium on Trial Readiness in Mitochondrial Myopathies. International Workshop:: Outcome measures and clinical trial readiness in primary mitochondrial myopathies in children and adults. Consensus recommendations. 16-18 November 2016, Rome, Italy. Neuromuscul Disord. 2017 Dec;27(12):1126-1137. doi: 10.1016/j.nmd.2017.08.006. Epub 2017 Sep 8. No abstract available. PMID 29074296
- [Background] Jung B, Martinez M, Claessens YE, Darmon M, Klouche K, Lautrette A, Levraut J, Maury E, Oberlin M, Terzi N, Viglino D, Yordanov Y, Claret PG, Bige N; Societe de Reanimation de Langue Francaise (SRLF); Societe Francaise de Medecine d'Urgence (SFMU). Diagnosis and management of metabolic acidosis: guidelines from a French expert panel. Ann Intensive Care. 2019 Aug 15;9(1):92. doi: 10.1186/s13613-019-0563-2. PMID 31418093
- [Background] Parikh S, Goldstein A, Koenig MK, Scaglia F, Enns GM, Saneto R, Anselm I, Cohen BH, Falk MJ, Greene C, Gropman AL, Haas R, Hirano M, Morgan P, Sims K, Tarnopolsky M, Van Hove JL, Wolfe L, DiMauro S. Diagnosis and management of mitochondrial disease: a consensus statement from the Mitochondrial Medicine Society. Genet Med. 2015 Sep;17(9):689-701. doi: 10.1038/gim.2014.177. Epub 2014 Dec 11. PMID 25503498
- [Background] Yang X, Xiao N, Yan J. The PedsQL in pediatric cerebral palsy: reliability and validity of the Chinese version pediatric quality of life inventory 4.0 generic core scales and 3.0 cerebral palsy module. Qual Life Res. 2011 Mar;20(2):243-52. doi: 10.1007/s11136-010-9751-0. Epub 2010 Sep 30. PMID 20882356
- [Background] Wong SS, Goraj B, Fung CW, Vister J, de Boer L, Koene S, Smeitink J. Radboud Centre for Mitochondrial Medicine Pediatric MRI score. Mitochondrion. 2017 Jan;32:36-41. doi: 10.1016/j.mito.2016.11.008. Epub 2016 Nov 16. PMID 27865797
- [Background] Panetta J, Smith LJ, Boneh A. Effect of high-dose vitamins, coenzyme Q and high-fat diet in paediatric patients with mitochondrial diseases. J Inherit Metab Dis. 2004;27(4):487-98. doi: 10.1023/B:BOLI.0000037354.66587.38. PMID 15303006
- See also: The detailed development, testing, manual and final version of International Paediatric Mitochondrial Disease Score (IPMDS) — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4987390/
- See also: Paediatric Quality of Life Inventory version 4.0 generic core scale (PedsQL 4.0 generic) — https://www.pedsql.org/
- See also: GRAS Notice, GRN No. 876. Hydroxytyrosol 2019 — https://www.fda.gov/media/134474/download